CLINICAL TRIAL: NCT03832751
Title: Estimation of Tissue Level of Human Beta-defensin 1 (HBD-1) in Vitiligo Before and After Narrowband UVB Phototherapy: a Case-control Study
Brief Title: Human Beta-defensin 1 in Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Fathy Elmasry, principal investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Dermatology 12
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitiligo patients (Experimental): Tissue levels of human beta-defensin 1 in vitiligo patients before and after NB-UVB phototherapy
  Interventions: Other: skin biopsy before and after NB-UVB phototherapy
- Healthy controls (Active Comparator): Tissue levels of human beta-defensin 1 in healthy controls
  Interventions: Other: skin biopsy before and after NB-UVB phototherapy

INTERVENTIONS:
Other: skin biopsy before and after NB-UVB phototherapy — skin biopsy before and after NB-UVB phototherapy to measure tissue human beta-defensin 1

SUMMARY:
There is a need to know the role of human beta defensin-1 in vitiligo pathogenesis and the probability of finding newer and effective therapy for vitiligo in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-segmental vitiligo.
* Both genders.
* Age more than 18 years old.
* New cases or cases not receiving any treatment for at least 3 months prior to the study.

Exclusion Criteria:

* Universal or segmental vitiligo.
* Any contraindication to phototherapy treatment.
* History of autoimmune diseases or other systemic diseases.
* Any other skin disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Tissue levels of human beta-defensin 1 before and after NB-UVB phototherapy | 6 months to 1 year